CLINICAL TRIAL: NCT05994170
Title: Reducing High Risk Primary Tumor Clinical Target Volumes (CTVp1) in Non-metastatic Nasopharyngeal Carcinoma Treated With Intensity-modulated Radiotherapy(IMRT): A Phase 3, Multicentre, Randomised Controlled Trial(CTVp1-NPC)
Brief Title: Reducing High Risk Primary Tumor Clinical Target Volumes (CTVp1) in Non-metastatic Nasopharyngeal Carcinoma
Acronym: CTVp1-NPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Collaborators: Sun Yat-sen University Cancer Centre (Unknown)
Responsible Party: Principal Investigator, Gui-Qiong Xu, Clinical Professor, Zhongshan People's Hospital, Guangdong, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSCPH-002
Record Dates: First submitted 2023-07-25; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Nasopharyngeal Carcinoma; Intensity-Modulated Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduction CTVp1 (Experimental): CTVp1=GTVp+5mm
  Interventions: Radiation: Reduction CTVp1
- Non-reduction CTVp1 (Placebo Comparator): CTVp1=GTVp+5mm+whole nasopharynx
  Interventions: Radiation: Non-reduction CTVp1

INTERVENTIONS:
Radiation: Reduction CTVp1 — High Risk Primary Tumor Clinical Target Volumes (CTVp1) is defined as 5mm margin from GTVp,including pre-induction chemotherapy tumor extension( CTVp1=GTVp+5mm)
  Arms: Reduction CTVp1
Radiation: Non-reduction CTVp1 — High Risk Primary Tumor Clinical Target Volumes (CTVp1) is defined as whole nasopharynx as well as 5mm margin from GTVp( CTVp1=GTVp+5mm+whole nasopharynx)
  Arms: Non-reduction CTVp1

SUMMARY:
To evaluate the long-term local control, survival rate, acute and late radiation related toxicities, quality of life after reducing high risk primary tumor clinical target volumes (CTVp1) in non-metastatic nasopharyngeal carcinoma treated with IMRT.

DETAILED DESCRIPTION:
This phase 3, multicenter,randomized controlled clinical trial recruits patients with newly-diagnosed non-metastatic nasopharyngeal carcinoma patients treated with IMRT. The intervention is delineating high risk primary tumor clinical target volumes (CTVp1) as GTV+5mm or GTV+5mm+whole nasopharynx. The objective is to compare the long-term local control, survival rate, acute and late radiation related toxicities between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. histologic confirmation of nonkeratinizing nasopharyngeal carcinoma(WHO II-III);
2. newly diagnosed stage I to IVa according to the American Joint Committee on Cancer-Union for International Cancer Control 8th edition stage-classification system
3. nasopharyngeal mass confined to one side of nasopharynx and did not exceed the midline(the line between the nasal septum and the midpoint of spinal cord/medulla) detected by electronic nasopharyngoscope (ENS) and magnetic resonance imaging (MRI). Pathological biopsy was recommended if it was unclear whether tumor invaded the contralateral side radiographically.
4. planned to receive curative IMRT, Chemotherapy drugs should be administered according to Chinese Society of Clinical Oncology (CSCO) guidelines depending on the TNM stage;(T1N0: No chemotherapy required;T2N0：No chemotherapy or concurrent cisplatin chemoradiotherapy if there are adverse prognostic indicators such as Epstein-Barr virus (EBV) DNA>4000 copies，node >3cm or with extranodal extension;T1-2N1: concurrent cisplatin chemoradiotherapy;T3N0: concurrent cisplatin chemoradiotherapy; stage III-Iva: platinum-based neoadjuvant chemotherapy+ concurrent cisplatin chemoradiotherapy+/-metronomic capecitabine therapy )
5. no previous treatment for cancer；
6. a Karnofsky performance-status score of at least 70 (on a scale from 0 to 100, with lower scores indicating greater disability);
7. between 18 and 70 years old;
8. adequate hematologic, renal, and hepatic function: Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;Adequate liver function: ALT and AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;Adequate renal function: BUN and CRE ≤ 1.5×ULN , endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
9. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. receipt of treatment with palliative intent;
2. receipt of previous treatment (radiotherapy, chemotherapy, or surgery [except diagnostic procedures]) to the nasopharynx;
3. had disease progress after neoadjuvant chemotherapy in local advantage NPC
4. presence of distant metastasis;
5. Keratinized squamous cell carcinoma or basal cell like squamous cell carcinoma;
6. Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
7. Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment;
8. lactation or pregnancy;
9. Any other condition including Mental disorder,drug or alcohol addition;do not have full capacity for civil acts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Local Relapse-free Survival(LRFS) | 3 years
  the time from randomization to documented local recurrence or death from any cause
Incidence of hearing impairment worse than graded 2 | 3 years
  audiometry and symptoms graded according to the CTCAE (version 5.0).

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  the time from randomization to documented death from any cause
Regional Relapse-free Survival(RRFS) | 3 years
  the time from randomization to documented regional recurrence or death from any cause
Distant metastasis-free survival (DMFS) | 3 years
  calculated from randomization to documented distant metastasis or death
Acute toxicities | 3 months
  Occur within 3 months after IMRT according Common Terminology Criteria for Adverse Events Version 5.0
Late toxicities | 3 years
  3 months after completion of radiotherapy graded according to both the Radiation Therapy Oncology Group criteria and the CTCAE (version 5.0)
Functional Assessment of Cancer Therapy-Head and Neck questionnaire (EORTC QLQ-H&N35) | 3 years
  Patient reported quality-of-life data and higher scores indicated more severe symptoms
Functional Assessment of Cancer Therapy-Head and Neck questionnaire (EORTC QLQ-C30) | 3 years
  Patient reported quality-of-life data and higher scores indicated more severe symptoms
radiation-induced otitis media with effusion (OME) | 3 years
  Evaluated by tympanometry
V60Gy | 3 years
  Volume that received at least 60Gy

CONTACTS AND LOCATIONS:
Overall Officials: Gui-qiong Xu, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China